CLINICAL TRIAL: NCT02816216
Title: Mobile Technology and Online Tools to Improve Asthma Control in Adolescents
Brief Title: Mobile Technology and Online Tools to Improve Asthma Control in Adolescents - Usability
Acronym: CampAir FEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: Columbia University (Other); New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R44HL127826 Usability; 5R44HL127826 (NIH)
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- End User Iterative Testing - CampAir (Other): To ensure the software and website function as intended, investigators will systematically test each of the seven CampAir modules with target end users. Participants will review one module per week for seven weeks. As part of each module, participants will also complete a daily asthma checklist. Following the review of each module, participants will be prompted to complete measures assessing technology acceptability and usability and product quality. Results will be used to modify and finalize the user interface and navigation to maximize usability.
  Interventions: Behavioral: CampAir

INTERVENTIONS:
Behavioral: CampAir — An empirically-based dynamic e-health intervention (based on the evidence-based ASMA) to assist adolescents with uncontrolled asthma to learn how to manage their illness and improve their asthma control.

SUMMARY:
This project will fully develop and preliminarily validate CampAir, an empirically-based dynamic e-health intervention (based on the evidence-based ASMA) to assist adolescents with uncontrolled asthma to learn how to manage their illness and improve their asthma control. In addition to developing a highly novel product for adolescents with asthma, the research proposed for this project will address unique scientific questions. Despite the high asthma prevalence among adolescents, few interventions have specifically targeted adolescents. This study is innovative in that it is among the few to focus on adolescents, who are often overlooked by the healthcare system. This research will assess factors associated with successful implementation of CampAir, thereby providing new information regarding how e-health interventions can be effectively developed and implemented for use with adolescents with asthma.

DETAILED DESCRIPTION:
This project will fully develop and preliminarily validate CampAir, an empirically-based dynamic e-health intervention (based on the evidence-based ASMA) to assist adolescents with uncontrolled asthma to learn how to manage their illness and improve their asthma control. In addition to developing a highly novel product for adolescents with asthma, the research proposed for this project will address unique scientific questions. Despite the high asthma prevalence among adolescents, few interventions have specifically targeted adolescents. This study is innovative in that it is among the few to focus on adolescents, who are often overlooked by the healthcare system. This research will assess factors associated with successful implementation of CampAir, thereby providing new information regarding how e-health interventions can be effectively developed and implemented for use with adolescents with asthma. To ensure the software and website function as intended, investigators will systematically test each of the seven CampAir modules with target end users. Participants will review one module per week for seven weeks. As part of each module, participants will also complete a daily asthma checklist. Following the review of each module, participants will be prompted to complete measures assessing technology acceptability and usability and product quality. Results will be used to modify and finalize the user interface and navigation to maximize usability. Results are expected to support that all participants find the CampAir product to be of high quality and technical acceptability. Participants are expected to rate the usability and relevance of the CampAir product highly. All participants are expected to advocate use of the product and recommend continued development and testing.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 13 - 18 years
* Prior Asthma diagnosis
* Use of a prescribed Asthma medication in the past 12 months

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
Product Evaluation | Once per module (One Evaluation per week for seven weeks)
  Participants will complete a brief online survey to rate the content modules and other components of the CampAir program in the areas of (a) engagement, (b) quality of content, (c) quality of flow, (d) value, (e) usefulness, (f) relevance to real-life, (g) usability. Open-ended questions will also be included to gather qualitative comments and recommendations for each area assessed. This measure will be repeated for each review with questions tailored to the particular components and modules reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Janey S McMillen, PhD, Principal Investigator — 3-C Institute for Social Development
Locations (1):
- 3-C Institute for Social Development, Durham, North Carolina, United States

REFERENCES:
- [Derived] Bruzzese JM, George M, Liu J, Evans D, Naar S, DeRosier ME, Thomas JM. The Development and Preliminary Impact of CAMP Air: A Web-based Asthma Intervention to Improve Asthma Among Adolescents. Patient Educ Couns. 2021 Apr;104(4):865-870. doi: 10.1016/j.pec.2020.09.011. Epub 2020 Sep 15. PMID 33004234